CLINICAL TRIAL: NCT01628042
Title: An Open-Label, Single-Dose Study to Investigate the Pharmacokinetics of MK-4618 in Patients With Renal Insufficiency
Brief Title: A Single Dose Study of the Pharmacokinetics of Vibegron (MK-4618) in Participants With Renal Insufficiency (MK-4618-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4618-014
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Participants With Severe Renal Insufficiency (Experimental): Participants will receive a single oral dose of vibegron 100 mg on Day 1.
  Interventions: Drug: Vibegron 100 mg
- Participants With Moderate Renal Insufficiency (Experimental): Participants will receive a single oral dose of vibegron 100 mg on Day 1.
  Interventions: Drug: Vibegron 100 mg
- Participants With Mild Renal Insufficiency (Experimental): Participants will receive a single oral dose of vibegron 100 mg on Day 1.
  Interventions: Drug: Vibegron 100 mg
- Healthy Matched Control Participants (Experimental): Participants receive a single oral dose of vibegron 100 mg on Day 1.
  Interventions: Drug: Vibegron 100 mg

INTERVENTIONS:
Drug: Vibegron 100 mg — Vibegron tablets, orally, on Day 1
  Other Names: MK-4618

SUMMARY:
This study will investigate the impact of impaired renal function on the plasma pharmacokinetics of vibegron (MK-4618) to guide use of vibegron in clinical trials in participants with overactive bladder and to guide recommendations on potential dosing adjustments for individuals with varying degrees of renal impairment.

ELIGIBILITY:
Inclusion Criteria - Renal Impaired Patients

* Body mass index (BMI) ≤40 kg/m^2
* Clinical diagnosis of renal insufficiency
* Stable baseline health

Inclusion Criteria - Healthy Subjects

- Stable baseline health

Exclusion Criteria - Renal Impaired Patients

* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, immunological, respiratory, or genitourinary disease
* History of recent stroke, chronic seizures, or major neurological disorder
* Demonstrated or suspected renal artery stenosis
* Renal transplant or nephrectomy
* History of cancer excepting certain skin or cervical cancers or cancers that were successfully treated 10 or more years prior to screening
* History of significant multiple and/or severe allergies (including latex allergy), or anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Unable to refrain from or anticipates the use of any medication including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of study drug, throughout the study, and until the post study visit
* Unable to avoid taking diuretics within 4 hours prior to dosing and 4 hours post dosing; must be on a stable dose for at least approximately 2 weeks (or 5 half-lives of the compound, whichever is longer)
* Unwilling to refrain from consuming any food or drink/beverage containing grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats 2 weeks prior to dosing until the post-study visit
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumption of excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Major surgery, donation or loss of 1 unit of blood (approximately 500 mL) within 4 weeks prior to administration of study drug
* Plasma donation within 7 days prior to administration of study drug
* Current regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months
* Nursing mother
* Participation in another investigational study within 4 weeks of study enrollment

Exclusion Criteria - Healthy Subjects

* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of stroke, chronic seizures, or major neurological disorder
* History of cancer excepting certain skin or cervical cancers or cancers that were successfully treated 10 or more years prior to screening
* History of significant multiple and/or severe allergies (including latex allergy), or anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Unable to refrain from or anticipates the use of any medication including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the dose of study drug, throughout the study, until the post study visit
* Unwilling to refrain from consuming any food or drink/beverage containing grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats 2 weeks prior to dosing until the post study visit
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumption of excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Major surgery, donation or loss of 1 unit of blood (approximately 500 mL) within 4 weeks prior to administration of study drug
* Plasma donation within 7 days prior to administration of study drug
* Current regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months
* Nursing mother
* Participation in another investigational study within 4 weeks of study enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2013-01-25 (Actual); Study Completion 2013-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Severe Renal Insufficiency; Participants With Moderate Renal Insufficiency; Participants With Mild Renal Insufficiency; Healthy Matched Control Participants: Participants received a single oral dose of vibegron 100 mg on Day 1.
Period: Overall Study
Arm/Group | Participants With Severe Renal Insufficiency | Participants With Moderate Renal Insufficiency | Participants With Mild Renal Insufficiency | Healthy Matched Control Participants
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Severe Renal Insufficiency | Participants With Moderate Renal Insufficiency | Participants With Mild Renal Insufficiency | Healthy Matched Control Participants | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Full Range); unit: Years] | 65 [53 to 75] | 64 [50 to 74] | 66 [59 to 75] | 57 [51 to 70] | 63 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC0-∞) After a Single Oral Dose of Vibegron 100 mg
Description: Blood samples were collected predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours after dosing in order to determine AUC0-∞ after a single oral dose of vibegron 100 mg.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: Per Protocol (PP) population, which included participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: nM•hr
Arm/Group | Participants With Severe Renal Insufficiency | Participants With Moderate Renal Insufficiency | Participants With Mild Renal Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8
nM•hr | 6337.17 [4940.96 to 8127.91] | 7137.53 [5615.70 to 9071.77] | 5156.07 [4045.44 to 6571.60] | 3466.04 [2663.08 to 4511.11]
Statistical Analysis 1: Comparison: Participants With Severe Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 1.83, 90% CI 2-sided [1.36 to 2.46]
Statistical Analysis 2: Comparison: Participants With Moderate Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 2.06, 90% CI 2-sided [1.55 to 2.74]
Statistical Analysis 3: Comparison: Participants With Mild Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 1.49, 90% CI 2-sided [1.11 to 2.00]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) After a Single Oral Dose of Vibegron 100 mg
Description: Blood samples were collected predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours after dosing in order to determine Cmax after a single oral dose of vibegron 100 mg.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: PP population, which included participants who complied with the protocol sufficiently to ensure that the data were likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Participants With Severe Renal Insufficiency | Participants With Moderate Renal Insufficiency | Participants With Mild Renal Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8
nM | 342.83 [232.00 to 506.62] | 404.50 [277.65 to 589.30] | 473.01 [323.26 to 692.12] | 240.80 [159.24 to 364.11]
Statistical Analysis 1: Comparison: Participants With Severe Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 1.42, 90% CI 2-sided [0.89 to 2.27]
Statistical Analysis 2: Comparison: Participants With Moderate Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ration = 1.68, 90% CI 2-sided [1.07 to 2.63]
Statistical Analysis 3: Comparison: Participants With Mild Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least-squares mean ratio = 1.96, 90% CI 2-sided [1.23 to 3.13]

3. Primary Outcome: Apparent Total Body Clearance (CL/F) After a Single Oral Dose of Vibegron 100 mg
Description: Blood samples were collected predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours after dosing in order to determine CL/F after a single oral dose of vibegron 100 mg.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 216, and 336 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Participants With Severe Renal Insufficiency | Participants With Moderate Renal Insufficiency | Participants With Mild Renal Insufficiency | Healthy Matched Control Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8
L/hr | 35.5 [27.68 to 45.53] | 31.5 [24.80 to 40.06] | 43.6 [34.23 to 55.61] | 64.9 [49.87 to 84.47]
Statistical Analysis 1: Comparison: Participants With Severe Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least squares mean ratio = 0.55, 90% CI 2-sided [0.41 to 0.74]
Statistical Analysis 2: Comparison: Participants With Moderate Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least squares mean ratio = 0.49, 90% CI 2-sided [0.36 to 0.65]
Statistical Analysis 3: Comparison: Participants With Mild Renal Insufficiency vs Healthy Matched Control Participants; Test type: Superiority or Other; ANCOVA; Geometric least squares mean ratio = 0.67, 90% CI 2-sided [0.50 to 0.90]

ADVERSE EVENTS:
Time Frame: Up to 336 hours post-dose
Description: The All Subjects as Treated (AST) population, which consisted of all participants who received at least 1 dose of the investigational drug, was used for the safety analysis.
Arm/Group | Participants With Severe Renal Insufficiency | Participants With Moderate Renal Insufficiency | Participants With Mild Renal Insufficiency | Healthy Matched Control Participants
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 4/8 | 3/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Participants With Severe Renal Insufficiency (N=8) | Participants With Moderate Renal Insufficiency (N=8) | Participants With Mild Renal Insufficiency (N=8) | Healthy Matched Control Participants (N=8)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0/0 (0) | 1/1 (1) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.